CLINICAL TRIAL: NCT03257111
Title: The Correlation Between Activity Levels and Rehabilitation Outcomes of Patients Post-stroke in an In-patient Rehabilitation Center
Brief Title: Activity Levels and Rehabilitation Outcomes of Patients Post-stroke
Status: Completed | Type: Observational
Sponsor: Florida Gulf Coast University (Other)
Collaborators: Brookdale Center for Healthy Aging & Rehabilitation (Unknown)
Responsible Party: Principal Investigator, Sherry Alexander, Research Compliance Coordinator, Florida Gulf Coast University
Other Study IDs: 2016-104
Record Dates: First submitted 2017-04-24; First posted 2017-08-22 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2018-02

CONDITIONS: Stroke
Keywords: rehabilitation outcomes; activity level
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: activity monitors — activity monitors are worn on the wrist, much like a watch. Data from the activity monitors will be downloaded once a week and at discharge. Normal hospital and therapy activities will not be altered.

SUMMARY:
Patients admitted to the in-patient rehabilitation center with a diagnosis of stroke will be recruited into the study. The participants will wear two activity monitors (one commercial grade and one research grade) for the duration of their rehab stay. Data from the monitors will be correlated with rehab outcomes, therapy units billed, and length of stay.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of stroke
* patient at the Brookdale Center for Healthy Aging & Rehabilitation
* not greater than maximum assistance to walk 10 feet
* walking re-training included in the therapy plan of care

Exclusion Criteria:

* primary diagnosis other than stroke
* allergy or reaction to the wrist bands of the activity monitors

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include only people with a diagnosis of stroke who have been admitted to the in-patient rehabilitation facility "Brookdale Center for Healthy Aging & Rehabilitation" in Naples, FL. The side of the stroke, the type of the stroke, or a history of prior stroke are not considerations. The study is intended to be very clinically focused to better understand the activity level of the population seen at the facility. This study is purposely not controlling the population to a very narrow presentation so that the results will speak directly to the facility and their outcomes
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2020-07-21 (Actual)

PRIMARY OUTCOMES:
Physical Activity Level | from the date of recruitment to the date of discharge or up to 45 days whichever comes first
  Amount of physical activity each day and throughout rehab stay as measured by 2 activity monitors beginning at admission and ending at discharge from the facility

SECONDARY OUTCOMES:
therapy units billed | from the date of recruitment to the date of discharge or up to 45 days whichever comes first
  therapy units are billed 15 minute time blocks; the number of each type of unit will be assessed at discharge from the facility
Functional Independence Measure (FIM) | from the date of recruitment to the date of discharge or up to 45 days whichever comes first
  FIM is a standard rehabilitation outcome used in all rehabilitation hospitals; measured at admission and discharge from the facility

CONTACTS AND LOCATIONS:
Overall Officials: Mollie Venglar, DSc, Principal Investigator — Florida Gulf Coast University
Locations (2):
- United States (2):
  - Florida Gulf Coast University, Fort Myers, Florida
  - Brookdale Center for Healthy Aging & Rehabilitation, Naples, Florida

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared outside of the research team